CLINICAL TRIAL: NCT00259246
Title: Fasting and Postprandial Response After Infusion of Saline, PYY1-36 and PYY3-36 and Effects on Appetite, Energy Intake and Energy Expenditure in Overweight/Obese Compared to Normalweight Subjects
Brief Title: The Role of Peptide YY (PYY)Infusions in Inhibiting Food Intake.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: EC-FP6 (contract number: LHM-CT-2003-503041) (Unknown); Aditech Pharma AB (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B208,1
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2005-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Drug: Peptide YY infusion

SUMMARY:
The aim of the study is to compare fasting and postprandial PYY levels between overweight/obese and lean subjects during and after an infusion of saline, PYY1-36 or PYY3-36 and to evaluate the efects on appetite, energy intake and energy expenditure.

DETAILED DESCRIPTION:
The study is a randomised dobbelblinded placebo controlled study with 24 male subjects ( 12 lean and 12 overweight/obese subjects). VAS scores are used to assess appetite and two ad libitum meals are served in the hours following the infusion. Energy expenditure is measured by ventilated hood system and blood is sampled during part of the study day.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI: 18-23 kg/m2) or 12 overweight/obese (BMI: 27-40 kg/m2)
* Body weight fluctuations < 5 kg over the past 2 months.
* Blood pressure normal to mildly hypertensive (<159/99 mm Hg)
* Non-elite athletes and not planning to change physical activity during the study.

Exclusion Criteria:

* Any physiological or psychological illnesses that could influence the study results
* Regular use of medicine
* Smoking defined as <1 cigarette per day.
* Substance abuse or dependence.
* Blood donation within the past 3 months before entering the study
* Drinking >21 alcoholic units/week.
* Food allergies.
* Special diets (e.g. vegetarian) or dislikes to any of the foods served during the study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2004-06; Study Completion 2005-11

PRIMARY OUTCOMES:
Appetite
Energy intake

SECONDARY OUTCOMES:
Energy expenditure and substrate oxidation
Blood parameters
Blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Principal Investigator — Department of Human Nutrition, RVAU